CLINICAL TRIAL: NCT04057001
Title: Hepatitis C Positive Organ to Recipient Hepatitis C Negative Longitudinal Transplant Study (HERCULES)
Brief Title: Hepatitis C Positive Organ to Recipient Hepatitis C Negative Longitudinal Transplant Study
Acronym: HERCULES
Status: Terminated | Type: Observational
Why Stopped: Unable to achieve adequate number of HCV+ donor offers
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000022932
Record Dates: First submitted 2019-06-13; First posted 2019-08-14 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Liver Transplant; Complications; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — RNA characterization of the tissue samples only. No plans for cell lines/ exome or genome sequencing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients who received a HCV+ liver transplant: Patients on a wait list for a liver transplant who agree to receiving a hepatitis C+ virus positive tested liver transplant.
- Patients who received a HCV- liver transplant: Patients on a wait list for a liver transplant who agree to receiving a hepatitis C- virus positive tested liver transplant.

SUMMARY:
Compare wait list mortality and time to liver, heart or kidney transplant for registrants listed to consider allografts from Hepatitis C Virus (HCV) Nucleic Amplification Testing (NAT)+ donors versus those who are not . The umbrella protocol has been set up to include heart and kidney transplant recipients.

DETAILED DESCRIPTION:
The research project will take place within each transplant center and can be incorporated into routine pre- and post-transplant care (i.e., no extra visits are needed). Enrolling in this study will enable patients to accept offers of HCV NAT+ livers, in addition to the regular waitlist. All other transplant eligibility criteria have to be met per routine care. The multi-site project will establish a biorepository and prospective data collection with the goal of obtaining more generalizable results than single-center studies alone can.

Patients who enroll in the study but receive an HCV- organ instead, will be (data collection only) as part of the study.

Aims are to evaluate sustained virologic response (SVR) rates post-transplant with Direct Acting Anti-Viral (DAA) therapy, as well as long-term patient and graft outcomes.

Evaluate the financial impact of timely transplant and DAA therapy compared to traditional wait time health care expenditure.

Create a blood and tissue biorepository for future evaluation of HCV NAT+ allografts and their outcomes

ELIGIBILITY:
Recipient Inclusion Criteria:

1. Adult patients > or = 18 years of age
2. Actively listed for Liver Transplant (LT) or Simultaneous Liver and Kidney (SLK)
3. Current HCV NAT- status
4. Review by multi-disciplinary transplant team that patient is appropriate for listing for HCV NAT+ liver offers

Recipient Exclusion Criteria:

1. Unwilling to consent to post transplant DAA therapy
2. Hepatitis B Virus (HBV) viremia

Donor Inclusion Criteria:

1. HCV NAT+
2. Deceased Donor organs
3. HBV cAb donors will be considered on a case by case basis based on specific recipient factors and plan for post-transplant prophylaxis

Donor Exclusion Criteria:

1. Bilirubin >3
2. Positive nucleotide testing for HBV
3. Radiographic, laboratory or other clinical evidence of portal hypertension
4. Fibrosis on pre-procurement liver biopsy fibrosis > F1 or fibroscan >7 (if both are done and discordant, use biopsy to determine eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients active on the waiting list for liver transplantation who are HCV NAT-
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Time to Transplant | 5 years
  Number of days between date of adding patient to the waitlist and transplant date comparing waitlist registrants listed to accept HCV NAT+ donor organs with those followed per standard of care (not accepting HCV NAT+ donor organs).

SECONDARY OUTCOMES:
Wait list Mortality | 5 years
  Number of days between adding patient to the waitlist to death on the waitlist comparing waitlist registrants listed to accept HCV NAT+ donor organs with those followed per standard of care (not accepting HCV NAT+ donor organs).

CONTACTS AND LOCATIONS:
Overall Officials: AnnMarie Liapakis, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States